CLINICAL TRIAL: NCT03522012
Title: Phase I, Double-Blind, Randomized, Three-Arm, Parallel-Group, Pharmacokinetic, Safety and Tolerability Study in Healthy Volunteers to Evaluate Bioequivalence of LusiNEX and Tocilizumab (EU and US)
Brief Title: Phase I, Pharmacokinetic, Safety and Tolerability Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mycenax Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LusiNEX-HV-PK-001
Record Dates: First submitted 2018-04-11; First posted 2018-05-11 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-11

CONDITIONS: Pharmacokinetics
Keywords: Pharmacokinetics; Tocilizumab
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- LusiNex (Experimental): 4 mg/kg, single-dose IV infusion (Mycenax tocilizumab)
  Interventions: Drug: Tocilizumab
- RoActemra (Active Comparator): 4 mg/kg, single-dose IV infusion (RoActemra; tocilizumab marketed in EU )
  Interventions: Drug: Tocilizumab
- Actemra (Active Comparator): 4 mg/kg, single-dose IV infusion (Actemra; tocilizumab marketed in US)
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab is a recombinant human monoclonal antibody of the immunoglobulin G1 subclass, directed against the IL-6 ligand specific receptor. By preventing the binding of IL-6 to its receptor, tocilizumab inhibits the biological activity of IL-6. Tocilizumab was approved by the US Food and Drug Administration (4 mg/kg with an increase to 8 mg/kg based upon clinical response) for the treatment of adult patients with moderate to severe active rheumatoid arthritis, who have had inadequate response to one or more tissue necrotizing factor (TNF) antagonist therapies. Tocilizumab is currently approved in 95 countries for the treatment of adult onset moderate to severe rheumatoid arthritis.
  Other Names: ACTEMRA

SUMMARY:
This is a randomized, double-blind, 3-arm, parallel-group single-dose study to compare the PK, PD, safety, tolerability, and immunogenicity of LusiNEX (Mycenax tocilizumab) versus RoActemra (EU tocilizumab) and Actemra (US tocilizumab) after a single IV infusion of 4 mg/kg in healthy volunteers (hereafter referred to as subjects). The therapeutic dose of tocilizumab starts with 4 mg/kg and ranges to 12 mg/kg, considering 4 mg/kg is the lowest dose, the same has been selected for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent prior to performing study-related procedures.
2. Healthy male or female aged between 18 to 55 years, inclusive.
3. A body mass index between 18 to 30 kg/m2, inclusive.
4. Medically healthy with clinically insignificant results (e.g., medical history, electrocardiograms [ECGs], and physical examination) as judged by the Principal Investigator at Screening/Day 1 (admission to study center).
5. All laboratory results including, but not restricted to, complete blood counts, liver function, and lipid profile should be within the normal range or clinically insignificant as judged by the Investigator at Screening/Day 1 (admission to study center). An abnormal laboratory result considered to be erroneous, may be repeated once during Screening at the discretion of the Investigator.
6. Have systolic blood pressure ≤140 and ≥90 mmHg, diastolic blood pressure ≤90 and ≥50 mmHg, and a heart rate ≥40 and ≤100 beats per minute at Screening/Day 1 (admission to study center).
7. Has to agree to abstain from alcohol intake 48 hours before administration of the study drug and during the inpatient period of the study.
8. Negative urine drug screen/alcohol breathylzer test at Screening/Day 1 (admission to study center).
9. Non-smokers or social smokers (defined as less than 10 cigarettes per week). No current use of any nicotine containing product. Cotinine levels ≤5 ng/mL.
10. Willing to abstain from sexual intercourse or use 2 methods of contraception (both male and female partners) as defined in the protocol for 3 months after study drug administration.

    Female subjects who are using oral hormonal contraceptives must be willing to use, with their partner, 2 methods of contraception as defined as defined in the protocol.
11. Has to agree to not donate sperm or ova for at least 3 months after study drug administration.
12. Subjects who are negative for hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibodies, human immunodeficiency virus I and II, as well as tuberculosis (TB) tests at Screening.
13. Did not receive a blood transfusion within 4 weeks prior to study drug administration, donate 400 mL or more blood within 8 weeks prior to study drug administration or donate plasma within 4 weeks prior to study drug administration and agrees to not make blood donations, including red blood cells, plasma, platelets, or whole blood for the duration of the study and for 3 months after study drug administration.
14. Able to be compliant with the protocol and attend all scheduled visits.
15. Has to agree to not consume any caffeine and/or xanthine products from 24 hours before admission to the study center until 48 hours after study drug administration.
16. Not have consumed grapefruit and/or grapefruit containing products, Seville oranges or quinine (tonic water) from 24 hours before admission to the study center until after the last sample has been collected for the study.

Exclusion Criteria:

1. Volunteers with any known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections.
2. Have been treated with IV antibiotics for an infection within 8 weeks or oral antibiotics within 2 weeks prior to Screening.
3. History of TB infection, active TB or latent TB infection, or recent exposure to a person with active TB.
4. Previous exposure to therapeutic monoclonal antibodies in the past 6 months prior to Screening.
5. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
6. A history of clinically significant gastrointestinal, renal, hepatic, cardiovascular, or allergic disease.
7. Evidence of active malignant disease, malignancies diagnosed within the previous 2 years (except basal cell carcinoma of the skin that has been excised and cured), or breast cancer diagnosed within the previous 2 years.
8. Impaired liver function as determined by:

   • Serum alanine aminotransferase and/or aspartate aminotransferase >1.5 x upper limit of normal (ULN) at Screening or admission to the study center. Subjects with values between ULN and 1.5 x ULN may be included in the study if considered not clinically significant by the Investigator.
9. Current or past history of diverticulitis or biliary obstruction.
10. Presence of proteinuria (other than trace amounts i.e., +, ++/+++) at Screening or admission to the study center.
11. Administration of an investigational product in another study within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to screening, or are currently participating in another clinical study of an investigational drug, or intending to participate in another clinical study of an investigational drug before completion of all scheduled evaluations in this clinical study.
12. Use of any prescription or over-the-counter medication (with the exception of contraceptive medication in females and paracetamol) within 7 days of Screening and for the duration of participation in the study. This includes the use of any NSAIDs (including aspirin) within 28 days before study drug administration and for the duration of participation in the study.
13. Intake of herbal drugs or dietary supplements excluding routine vitamins but including megadose (intake of 20 to 600 times the recommended daily dose) vitamin therapy within 28 days prior to study drug administration, unless agreed as not clinically relevant by the Investigator and Sponsor.
14. Regular alcohol consumption of >14 (female subjects) or >21 (male subjects) units of alcohol per week at the time of Screening (1 unit = 150 mL of wine or 360 mL of beer or 45 mL of 40% alcohol).
15. Failure to satisfy the Principal Investigator of fitness to participate for any other reason.
16. Female subjects who are pregnant, trying to become pregnant, or lactating.
17. Subjects who have a history of relevant drug hypersensitivity or hypersensitivity to the active substance or to any of the excipients.
18. Inability to undergo venipuncture and/or tolerate venous access.
19. Subjects who do not agree to use medically acceptable methods of contraception (as defined in the protocol).
20. Involvement in the planning and/or conduct of the study (applies to the Sponsor, Contract Research Organizations, and study center staff, etc.).
21. Subjects who are unlikely to co-operate with the requirements of the study.
22. Any live virus vaccination or planned vaccination within 28 days before Screening and for the duration of participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 2 months
  Area under concentration-time curve from time 0 (predose) extrapolated to infinity (AUC(0-∞)).

SECONDARY OUTCOMES:
Cmax | 2 months
  Maximum concentration (Cmax)
tmax | 2 months
  Time to reach maximum concentration (tmax)
AUC(0-t) | 2 months
  Area under concentration-time curve from time 0 (predose) to the last quantifiable data point (AUC(0-t))
t1/2 | 2 months
  Terminal half-life (t1/2)
Vss | 2 months
  Volume of distribution at steady-state
Vd | 2 months
  Volume of distribution (Vd)
CL | 2 months
  Systemic clearance (CL)
Kel | 2 months
  Elimination rate constant (Kel)
AEs | 2 months
  The Investigator will carefully monitor each subject throughout the study for any AEs (coded to preferred term and system organ class using the Medical Dictionary for Regulatory Activities [MedDRA])
antidrug antibodies | 2 months
  means of the occurrence of antidrug antibodies (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Walsh, Dr., Principal Investigator — Nucleus Network Ltd
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia